CLINICAL TRIAL: NCT03639792
Title: Escorting Octogenarian for Gastric Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, BIRENDRA KUMAR SAH, Surgeon, Ruijin Hospital
Other Study IDs: RJ-GC-Postop-complication 2
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2018-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; postoperative complication; octogenarian
MeSH Terms: conditions — Stomach Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: gastric cancer surgery — Gastric cancer surgery

SUMMARY:
An objective analysis of postoperative complications is vital to escort octogenarian for gastric cancer surgery. Investigator carefully collected clinical data prospectively to pave way for standard management in high risk patients.

DETAILED DESCRIPTION:
An objective analysis of postoperative complications is vital to escort octogenarian for gastric cancer surgery. Investigator carefully collected clinical data prospectively to pave way for standard management in high risk patients. Detailed data on surgical indication, assessment for proposed surgery and perioperative management are analyzed for future guidelines in senile.

ELIGIBILITY:
Inclusion Criteria:

- Pathologically confirmed gastric cancer patients Clinically fit for gastric cancer surgery

Exclusion Criteria:

- Non gastric cancer patients Clinically unfit for gastric cancer surgery

Ages: 80 Years to 90 Years | Sex: All
Age Groups: Older Adult
Study Population: A cohort of gastric cancer patients who underwent surgery during two consecutive years in a Chinese hospital.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Morbidity and mortality | One month after hospital discharge
  Postoperative Morbidity and mortality according to standard definition

SECONDARY OUTCOMES:
Overall survival | upto two years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Birendra K Sah, Ph D, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China